CLINICAL TRIAL: NCT02531490
Title: Personalized Hemodynamically Guided Antihypertensive Treatment in Pregnant Women With Mild to Moderate Hypertension: a Randomized Controlled Trial
Brief Title: Early Vascular Adjustments During Hypertensive Pregnancy
Acronym: EVA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: METC152017
Record Dates: First submitted 2015-08-05; First posted 2015-08-24 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Hypertension, Pregnancy-Induced; Pre-Eclampsia
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — Labetalol; Nifedipine; Methyldopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- randomized, interventiongroup (Active Comparator): Women with a hyperdynamic vasodilated profile, characterized by a mean arterial pressure (MAP)/ Heart rate (Hr) ratio ≤ 1.1 are prescribed a beta-blocker. Women with a hypodynamic vasoconstrictive profile (MAP/Hr ratio ≥ 1.4) are prescribed nifedipine. Women with normodynamic profile (MAP/Hr ratio in between 1.1 and 1.4) are prescribed Methyldopa.
  Interventions: Drug: Labetalol; Drug: Nifedipine; Drug: Methyldopa
- randomized, control-group (No Intervention): Women who give informed consent for randomization, and are randomized to the control group will not be medicinally treated for mild to moderate gestational hypertension.
- not-randomized, control-group (No Intervention): Women who do not want to be randomized, but who give informed consent for follow-up on their data until discharge after delivery. They will receive standard care, i.e. no medication is prescribed for mild to moderate gestational hypertension.

INTERVENTIONS:
Drug: Labetalol
  Other Names: Trandate
  Arms: randomized, interventiongroup
Drug: Nifedipine
  Other Names: Adalat
  Arms: randomized, interventiongroup
Drug: Methyldopa
  Other Names: Aldomet
  Arms: randomized, interventiongroup

SUMMARY:
Paradoxical fetal and maternal results of studies have led to inconsistent use of antihypertensive drugs or no treatment at all in mild to moderate gestational hypertension in the Netherlands. However, none of the studies have taken the individual maternal circulatory state or the contemplated blood pressure response into account. Hypertension may be accompanied by high (hyperdynamic vasodilated profile), normal (normodynamic profile) of low (hypodynamic vasoconstrictive profile) cardiac output, and preeclampsia is not restricted to one circulatory profile. Therefore antihypertensive drugs should be viewed upon as correctors of the hemodynamic state rather than solely reducers of blood pressure. Without taking the maternal hemodynamic profile and condition into account, generic antihypertensive treatment can be expected to result in disappointing, inadequate and paradoxical results. The investigators hypothesize that in mild to moderate hypertension, personalized hemodynamically guided antihypertensive therapy (with target systolic and diastolic blood pressure <130/80mmHg), prevents the progression to severe hypertension and/or preeclampsia compared to no treatment, without the alleged side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18years or older
* Before 37 weeks of gestational age;
* Diagnosed with mild to moderate gestational hypertension

Exclusion Criteria:

* Women with severe hypertension: systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 110mmHg.
* Women with chronic hypertension who are already on antihypertensive drugs. If no antihypertensive drugs are used yet, women with pre-existent hypertension are eligible to participate.
* Women diagnosed with preeclampsia or eclampsia in the current pregnancy.
* Women who are not able to comprehend the study outline.
* Women who have already participated in this study cannot be included a second time.
* Women who have a (relative) contra-indication for one of the possible prescribed medications (for example women who have tested positive for antinuclear antibodies, which is a contraindication for Methyldopa).
* Women who intend to terminate the pregnancy
* Women who have a fetus with a major anomaly or chromosomal abnormality

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 368 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
number of patients with severe gestational hypertension | from date of randomization until the date of this study event, assessed up to 1 week post partum (maximum 23weeks after inclusion)
  Systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 110mmHg, measured at every visit
number of patients with preeclampsia | from date of randomization until the date of this study event, assessed up to 1 week post partum (maximum 23weeks after inclusion)
  Preeclampsia is defined as the coexistence of de novo hypertension after 20 weeks of gestation and one or more of the following new-onset conditions:
  1. Proteinuria (spot urine protein/creatinine ≥ 30g/mol or ≥ 300mg/day or at least 1 g/L [2+] on dipstick testing).
  2. Other maternal organ dysfunction:
     * Renal insufficiency (creatinine levels ≥ 90μmol/L);
     * Liver involvement (elevated transaminases: ASAT ≥31 U/L and/or ALAT ≥34U/L);
     * Neurological complications (hyperreflexia when accompanied by clonus and/or severe headaches, persistent visual scotomata, altered mental status, eclampsia);
     * Haematological complications (thrombocytopenia, platelet count below 150.000/dL, disseminated intravascular coagulation, haemolysis).

SECONDARY OUTCOMES:
the pattern of change of the hemodynamic profile, measured by the ratio of mean arterial pressure and heart rate. | at baseline and each study visit/follow up measurement (at 1 week, 2 weeks, etc. up to 23 weeks after inclusion. The expected average is 8 weeks
  hemodynamic profiles will be classified as hyperdynamic, hypodynamic vasocontricted or mixed profile.
hemodynamic profile by mean arterial pressure/heart rate ratio | from date of randomization until the date of study event, assessed up to 1 week post partum (maximum 23weeks after inclusion)
  hemodynamic profiles will be classified as hyperdynamic, hypodynamic vasocontricted or mixed profile.
diameter aortic outflow tract and left ventricular outflow tract measured by transthoracic echocardiography | from baseline, and every 4 weeks (maximum 6 times, because in max. 23 weeks end of study is reached)
  cardiac output can be derived from these values + heart rate
left ventricular volume after diastole and systole measured by transthoracic echocardiography | from baseline, and every 4 weeks (maximum 6 times, because in max. 23 weeks end of study is reached)
  ejection fraction can be derived from these values
diameter aortic outflow tract and left ventricular outflow tract measured by transthoracic echocardiography | from date of randomization until the date of study event, assessed up to 1 week post partum (maximum 23weeks after inclusion)
  cardiac output can be derived from these values + heart rate
left ventricular volume after diastole and systole measured by transthoracic echocardiography | from date of randomization until the date of study event, assessed up to 1 week post partum (maximum 23weeks after inclusion)
  ejection fraction can be derived from these values
cardiac remodeling during pregnancy: number of patients with concentric left ventricular remodeling or concentric hypertrophy. | from baseline, and every 4 weeks (maximum 6 times, because in max. 23 weeks end of study is reached)
  Echocardiographic concentric left ventricular (LV) remodelling and hypertrophy. Concentric remodeling is defined as a relative wall thickness (RWT) <=0.43 with a Left Ventricular Mass index (LVMi) of <95 gram/m2. Concentric hypertrophy is defined as a RWT <0.43 with a LVMi of ≥95 gram/m2.
cardiac remodeling during pregnancy: number of patients with concentric left ventricular remodeling or concentric hypertrophy. | from date of randomization until the date of study event, assessed up to 1 week post partum (maximum 23weeks after inclusion)
  Echocardiographic concentric left ventricular (LV) remodelling and hypertrophy. Concentric remodeling is defined as a relative wall thickness (RWT) <=0.43 with a Left Ventricular Mass index (LVMi) of <95 gram/m2. Concentric hypertrophy is defined as a RWT <0.43 with a LVMi of ≥95 gram/m2.
health status of the newborn by Apgar score | assessed immediately after delivery
  scored by gynecologist or paediatrician on a scale of 1 to 10
prevalence of small for gestational age infancy | assessed at delivery date
  birth weight and percentile combined with gestational age at delivery
prevalence of premature neonates | assessed at delivery date
  gestational age at delivery
number of a composite of adverse neonatal outcomes | from delivery up neonates will be followed for the duration of the hospital stay, an expected average of 6 weeks
  Stillbirth, perinatal mortality, morbidity: chronic lung disease, neonatal sepsis, severe intra-ventricular haemorrhage (IVH) > grade II, periventricular leucomalacia > grade I, and necrotizing enterocolitis. Days on ventilation support, length of admission in neonatal intensive care, and total days in hospital until 3 months corrected age.
maternal well-being questionnaire, | at baseline and each study visit/follow up measurement (at 1 week, 2 weeks, etc. up to 23 weeks after inclusion. The expected average is 8 weeks
  Reported medication side effects, and maternal well-being by signs and symptoms during pregnancy
number of assessed maternal complications | from a study event participants will be followed for the duration of hospital stay, an expected average of 1 week
  Composite of maternal complications including: mortality, stroke, eclampsia, blindness, uncontrolled hypertension, respiratory failure, birth related variables, needed level of care
gestational age at the moment of progression to primary outcome. | from baseline/inclusion until a study event is reached (up to 18 weeks after inclusion), with an expected average of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Spaanderman, professor, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

REFERENCES:
- [Background] Schutte JM, Schuitemaker NW, van Roosmalen J, Steegers EA; Dutch Maternal Mortality Committee. Substandard care in maternal mortality due to hypertensive disease in pregnancy in the Netherlands. BJOG. 2008 May;115(6):732-6. doi: 10.1111/j.1471-0528.2008.01702.x. PMID 18410657
- [Background] Abalos E, Duley L, Steyn DW. Antihypertensive drug therapy for mild to moderate hypertension during pregnancy. Cochrane Database Syst Rev. 2014 Feb 6;(2):CD002252. doi: 10.1002/14651858.CD002252.pub3. PMID 24504933
- [Background] Easterling TR, Benedetti TJ, Schmucker BC, Millard SP. Maternal hemodynamics in normal and preeclamptic pregnancies: a longitudinal study. Obstet Gynecol. 1990 Dec;76(6):1061-9. PMID 2234714
- [Background] Valensise H, Vasapollo B, Gagliardi G, Novelli GP. Early and late preeclampsia: two different maternal hemodynamic states in the latent phase of the disease. Hypertension. 2008 Nov;52(5):873-80. doi: 10.1161/HYPERTENSIONAHA.108.117358. Epub 2008 Sep 29. PMID 18824660
- [Background] Taler SJ, Textor SC, Augustine JE. Resistant hypertension: comparing hemodynamic management to specialist care. Hypertension. 2002 May;39(5):982-8. doi: 10.1161/01.hyp.0000016176.16042.2f. PMID 12019280
- [Derived] Mulder E, Ghossein-Doha C, Appelman E, van Kuijk S, Smits L, van der Zanden R, van Drongelen J, Spaanderman M. Study protocol for the randomized controlled EVA (early vascular adjustments) trial: tailored treatment of mild hypertension in pregnancy to prevent severe hypertension and preeclampsia. BMC Pregnancy Childbirth. 2020 Dec 12;20(1):775. doi: 10.1186/s12884-020-03475-w. PMID 33308198